CLINICAL TRIAL: NCT02997215
Title: Effect of Intravenous Lidocaine on Postoperative Pain Management After Laparoscopy Cholecystectomy
Brief Title: Intravenous Lidocaine and Postoperative Pain Management
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, YANXIA SUN, Vice-Chief Anesthesiologist, Beijing Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-YJJ-GGL-008
Record Dates: First submitted 2016-12-06; First posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Postoperative Pain Management
Keywords: intravenous lidocaine; postoperative pain management
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intravenous lidocaine (Experimental): intravenous lidocaine 1.5mg/kg during induction then infused at 2mg/kg/h until the end of procedure.
  Interventions: Drug: Lidocaine
- saline placebo (Placebo Comparator): same amount volume saline infusion
  Interventions: Drug: Saline Placebo

INTERVENTIONS:
Drug: Lidocaine — lidocaine infusion during surgery
  Arms: intravenous lidocaine
Drug: Saline Placebo — saline infusion at same rate as intervention group during surgery
  Arms: saline placebo

SUMMARY:
This study was to evaluate the effect of intraoperative intravenous lidocaine on postoperative pain management after laparoscopic cholecystectomy. Half of patients will receive intravenous lidocaine during procedure, the rest half of patients will receive regular anesthesia care and placebo treatment.

DETAILED DESCRIPTION:
Postoperative pain and ileus are primary reasons for delayed patient recovery and longer hospital stays after abdominal surgery. Opioids have been widely used to treat pain in this patient population. However, opioid administration can exacerbate postoperative ileus and further delay patient recovery. Multimodal approaches and adjunctive therapies are therefore recommended for pain control after abdominal surgery to reduce opioid consumption and opioid-related adverse effects.

Studies have reported that systemically administered lidocaine has analgesic, anti-inflammatory, and anti-hyperalgesic effects. Several clinical trials have been published that evaluated systemically administered lidocaine for postoperative pain management and recovery after surgery. However, the evidence for beneficial effects of systemic lidocaine for postoperative recovery remains controversial. Therefore, the investigators performed this study to evaluate the efficacy of systemic administration of lidocaine for postoperative analgesia and gastrointestinal recovery after laparoscopic cholecystectomy. The investigators primary hypothesis is that systemic lidocaine administration reduces pain intensity following surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) status I-II adult patients undergoing elective laparoscopic cholecystectomy.

Exclusion Criteria:

* Open surgery;
* Patients allergic to lidocaine or other local anesthetics;
* Drug abuser.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
postoperative pain score | 6 hours after surgery
  visual analogue score (1-10)
postoperative pain score | 24 hours after surgery
  visual analogue score (1-10)
postoperative pain score | 72 hours after surgery
  visual analogue score (1-10)
total postoperative opioid consumption | 48 hours after surgery
  postoperative fentanyl consumption

SECONDARY OUTCOMES:
incidence of postoperative complication | 48 hours after surgery
  opioid-related side effects, such as nausea and vomiting, and the incidence of adverse effects associated with systemic administration of lidocaine.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology; Beijing Tongren Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participants data for primary and secondary outcome measures will be available within 6 months of study completion